CLINICAL TRIAL: NCT07387536
Title: The Effectiveness of Topical Silicone Application Combined With Photoprotection in the Development of Scarring Following Blepharoplasty
Acronym: ETSACPDSFP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEI-2025/05/05
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Scar Formation
Keywords: Upper Blepharoplasty Approach; Post-operative Scar; Vancouver Scar Scale
MeSH Terms: interventions — Sunscreening Agents

STUDY DESIGN:
Intervention Model Description: Improscar Stick® 50, a silicone-based topical formulation with sunscreen (SPF 50), will be administered to the eyelid incisions of research participants who have undergone blepharoplasty. The treatment protocol will commence in the first postoperative week and will be prescribed for application twice daily for a minimum duration of three months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Improscar Stick® 50, a silicone-based topical formulation with sunscreen (SPF 50) application (Experimental)
  Interventions: Drug: Silicone-based topical formulation with sunscreen (SPF 50) application

INTERVENTIONS:
Drug: Silicone-based topical formulation with sunscreen (SPF 50) application — Silicone-based topical formulation with sunscreen (SPF 50), will be administered to the eyelid incisions of research participants who have undergone blepharoplasty.

SUMMARY:
Assess the efficacy of utilizing topical silicone with photoprotection (Improscar Stick® 50) on the quality of healing following upper blepharoplasty, employing the Vancouver and POSAS scales (both patient and observer) over a minimum follow-up period of three months.

DETAILED DESCRIPTION:
This study is a clinical, experimental, prospective, and comparative before-and-after investigation involving participants undergoing upper blepharoplasty. Individuals aged between 18 and 70 years will be included in the study. Clinical assessments will be conducted at four distinct time points: one week postoperatively (coinciding with suture removal and the initiation of treatment), one week following the commencement of treatment, at one month, and three months post-treatment. The Vancouver and POSAS scales, both subjective and objective, will be employed for evaluation. For inferential analysis, ANOVA for repeated measures will be utilized, employing IBM SPSS Statistics v31.0 software. Any adverse effects will be documented.

ELIGIBILITY:
Inclusion Criteria:

* The study participants are individuals aged 18 years and older, encompassing both male and female subjects. These participants are undergoing blepharoplasty and have provided their written informed consent to partake in the research.

Exclusion Criteria:

* Individuals with a history of previous surgical procedures on the eyelids, apart from the current blepharoplasty. . Those who have previously undergone intralesional modulation are also considered. Individuals with a known allergy to any components of the product under investigation. The presence of local skin infections in the treatment area. Suspicious skin lesions suggestive of malignancy in the eyelid region. Pregnancy or breastfeeding during the study. - Research subjects who, after being included in the study, do not complete the scheduled clinical follow-up. Research subjects who discontinue the use of the topical treatment before the end of the established period. Voluntary withdrawal of informed consent at any stage of the study. Later detection of exclusion criteria that were not identified during the initial evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Objetive evaluation | From enrollment to the end of treatment at 3 months
  To objectively evaluate the quality of post-surgical eyelid scars, assessments will be conducted based on the Vancouver scale, focusing on vascularity, pigmentation, pliability, and height.
Subjective evaluation | From enrollment to the end of treatment at 3 months
  For subjective evaluation, the POSAS scale will be employed, which consists of two components: one completed by the research subject and the other by the clinical observer. Each component assesses six domains-color, thickness, relief, itching, and pain-using a scoring system ranging from 1 (normal skin) to 10 (worst possible outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oftalmologia F.A.P. Conde de Valenciana, I.A.P., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From march to December 2026

REFERENCES:
- [Result] Chen L, Hu JY, Wang SQ. The role of antioxidants in photoprotection: a critical review. J Am Acad Dermatol. 2012 Nov;67(5):1013-24. doi: 10.1016/j.jaad.2012.02.009. Epub 2012 Mar 9. PMID 22406231
- [Result] Zhang B, Yang E, Zhang H. Efficacy of Early Application of 1540 nm Non-ablative Fractional Laser and Silicones to Improve Post-epicanthoplasty Scars. Aesthetic Plast Surg. 2022 Oct;46(5):2452-2458. doi: 10.1007/s00266-022-02866-y. Epub 2022 Apr 1. PMID 35364722
- [Result] Karanfilian TS, Thuma T, Cheng T, Paramo R, Moon JY, Akella S, Barmettler A. Efficacy of Silicone Gel Versus Placebo for Postsurgical Scars of the Eyelids: A Randomized, Controlled, Double-Blinded Study. Ophthalmic Plast Reconstr Surg. 2025 Sep-Oct 01;41(5):555-559. doi: 10.1097/IOP.0000000000002913. Epub 2025 Feb 13. PMID 39946309
- [Result] Quinn KJ, Evans JH, Courtney JM, Gaylor JD, Reid WH. Non-pressure treatment of hypertrophic scars. Burns Incl Therm Inj. 1985 Dec;12(2):102-8. doi: 10.1016/0305-4179(85)90035-x. PMID 4092154
- [Result] Chang CC, Kuo YF, Chiu HC, Lee JL, Wong TW, Jee SH. Hydration, not silicone, modulates the effects of keratinocytes on fibroblasts. J Surg Res. 1995 Dec;59(6):705-11. doi: 10.1006/jsre.1995.1227. PMID 8538169
- [Result] Bleasdale B, Finnegan S, Murray K, Kelly S, Percival SL. The Use of Silicone Adhesives for Scar Reduction. Adv Wound Care (New Rochelle). 2015 Jul 1;4(7):422-430. doi: 10.1089/wound.2015.0625. PMID 26155385
- [Result] Monstrey S, Middelkoop E, Vranckx JJ, Bassetto F, Ziegler UE, Meaume S, Teot L. Updated scar management practical guidelines: non-invasive and invasive measures. J Plast Reconstr Aesthet Surg. 2014 Aug;67(8):1017-25. doi: 10.1016/j.bjps.2014.04.011. Epub 2014 May 14. PMID 24888226
- [Result] Tran B, Wu JJ, Ratner D, Han G. Topical Scar Treatment Products for Wounds: A Systematic Review. Dermatol Surg. 2020 Dec;46(12):1564-1571. doi: 10.1097/DSS.0000000000002712. PMID 32932267
- [Result] Stavrou D, Weissman O, Winkler E, Yankelson L, Millet E, Mushin OP, Liran A, Haik J. Silicone-based scar therapy: a review of the literature. Aesthetic Plast Surg. 2010 Oct;34(5):646-51. doi: 10.1007/s00266-010-9496-8. Epub 2010 Mar 31. PMID 20354695
- [Result] Guclu ES, Ozer O, Celik S, Eroz P, Baysal Z. Comparison of the Cosmetic Efficacy of Extractum Cepae and Silicone-Based Gel in Upper Blepharoplasty. J Craniofac Surg. 2024 Oct 1;35(7):e658-e660. doi: 10.1097/SCS.0000000000010472. Epub 2024 Jul 17. PMID 39016346
- [Result] Eilers RE Jr, Ross EV, Cohen JL, Ortiz AE. A Combination Approach to Surgical Scars. Dermatol Surg. 2016 May;42 Suppl 2:S150-6. doi: 10.1097/DSS.0000000000000750. PMID 27128241
- [Result] Gupta S, Kalra A. Efficacy and safety of intralesional 5-fluorouracil in the treatment of keloids. Dermatology. 2002;204(2):130-2. doi: 10.1159/000051830. PMID 11937738
- [Result] Kerwin LY, El Tal AK, Stiff MA, Fakhouri TM. Scar prevention and remodeling: a review of the medical, surgical, topical and light treatment approaches. Int J Dermatol. 2014 Aug;53(8):922-36. doi: 10.1111/ijd.12436. Epub 2014 Apr 2. PMID 24697346
- [Result] Kalasho BD, Kikuchi R, Zoumalan CI. Silicone-Based Scar Cream for Post Upper Eyelid Blepharoplasty-associated Cicatricial and Hypertrophic Scarring. J Drugs Dermatol. 2019 May 1;18(5):440-446. PMID 31141848
- [Result] Drolet BC, Sullivan PK. Evidence-based medicine: Blepharoplasty. Plast Reconstr Surg. 2014 May;133(5):1195-1205. doi: 10.1097/PRS.0000000000000087. PMID 24776550